CLINICAL TRIAL: NCT01896154
Title: A Randomized, Controlled Clinical Study on the Effect of Non-digestible Polysaccharides (NPS) on the Immune Response to Influenza Vaccination in Elderly
Brief Title: Pilot Study on Effect Size of Non-digestible Polysaccharides (NPS) on Immunity
Acronym: Fib-P-2012
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: European Commission (Other); Food & Biobased Research - Wageningen UR (Unknown); Teagasc (Industry); Nofima (Other); BioActor B.V. (Industry); Swedish Oat Fiber AB (Unknown); Immitec (Unknown); Institut Pasteur (Industry); University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Fib-P-2012
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2015-02

CONDITIONS: Immunosenescence
Keywords: dietary fibers, influenza vaccination, HI titres
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- NPS from yeast (Experimental): Powder containing the active ingredients (500mg NPS from yeast) as well as filling substances (maltodextrins) and flavour adding up to 12.0 g altogether in sachets; consumed once daily after having been stirred in milk or filtered apple juice (ca. 200 ml/ 1 glass) for 5 weeks. 2 weeks before vaccination and 3 weeks after vaccination.
  Interventions: Dietary Supplement: NPS
- NPS from shiitake (Experimental): Powder containing the active ingredient (500mg NPS from shitake) as well as filling substances (maltodextrins) and flavour adding up to 12.0 g altogether in sachets; consumed once daily after having been stirred in milk or filtered apple juice (ca. 200 ml/ 1 glass) for 5 weeks: 2 weeks before vaccination and 3 weeks after vaccination.
  Interventions: Dietary Supplement: NPS
- NPS from oat (Experimental): Powder containing the active ingredient (10g NPS from oat) as well as filling substances (maltodextrins) and flavour adding up to 12.0 g altogether in sachets; consumed once daily after having been stirred in milk or filtered apple juice (ca. 200 ml/ 1 glass) for 5 weeks: 2 weeks before vaccination and 3 weeks after vaccination.
  Interventions: Dietary Supplement: NPS
- NPS from wheat (Experimental): Powder containing the active ingredient (10g NPS from wheat) as well as filling substances (maltodextrins) and flavour adding up to 12.0 g altogether in sachets; consumed once daily after having been stirred in milk or filtered apple juice (ca. 200 ml/ 1 glass) for 5 weeks: 2 weeks before vaccination and 3 weeks after vaccination.
  Interventions: Dietary Supplement: NPS
- NPS from Lactobacillus mucosae (Experimental): Powder containing the active ingredient (2,3g NPS from L. mucosae) as well as filling substances (maltodextrins) and flavour adding up to 12.0 g altogether in sachets; consumed once daily after having been stirred in milk or filtered apple juice (ca. 200 ml/ 1 glass) for 5 weeks: 2 weeks before vaccination and 3 weeks after vaccination.
  Interventions: Dietary Supplement: NPS
- Maltodextrin (Placebo Comparator): 12.0 g Maltodextrin and flavour with identical/similar appearance and taste (when mixed in drink), consumed once daily as described for the active products (NPS.
  Interventions: Dietary Supplement: NPS

INTERVENTIONS:
Dietary Supplement: NPS — Comparison of multiple dietary non-digestible polysaccharides

SUMMARY:
The aim of the study is to estimate the effect size of a 5-week consumption period of different dietary non-digestible polysaccharides (NPS) on antibody response to influenza vaccination and cellular immunity of healthy volunteers (aged ≥ 50) for clarifying whether these NPS may enable enhancement of immune defence and to estimate the sample size for a confirmative trial. Furthermore the effects on faecal microbiota and its metabolites will be investigated.

DETAILED DESCRIPTION:
The study is conducted in the frame of the collaborative project 'FibeBiotics' (Nr. 289517) (Fibers as support of the Gut and Immune function of Elderly - From polysaccharide compound to health claim) within the Seventh Framework Programme (FP7) for Research and Technological Development of the European Union (EU).

ELIGIBILITY:
Inclusion Criteria:

* Free-living postmenopausal woman and men aged ≥ 50 years willing to have influenza vaccination season 2012/2013
* willingness to abstain as far as possible from food and supplements containing probiotics, prebiotic supplements, other fermented products, supplements containing vitamins and minerals as well as willing to sustain on a low dietary fibre diet for 7 weeks.
* written informed consent

Exclusion Criteria:

* Subjects enrolled in another clinical study in the last 4 weeks
* Subjects already vaccinated against influenza during 2012-2013 with either the influenza vaccine used in the present study or another influenza vaccine
* vaccination against influenza within the previous 10 months
* suffering from influenza or influenza-like illness within the previous 10 months
* other vaccinations during and within 2 months before the study
* symptoms of common infectious diseases (CID) of the airways or other organ systems e.g. gastrointestinal tract in the last 4 weeks before inclusion
* known congenital, acquired or iatrogenic immunodeficiency (e.g. HIV, chemotherapy, immunosuppression)
* active autoimmune diseases
* allergy or hypersensitivity to any component of the vaccine (e. g. chicken egg protein, certain antibiotics)(s. a. 9.2)
* allergy or hypersensitivity to any component of the test product (e. g. yeast, gluten, shiitake mushrooms)
* allergy to latex
* known coeliac disease (gluten enteropathy)
* bowel movement less than 3 times per week
* subjects, who meet 2 or more Rome III criteria for constipation or who take laxatives on a regular basis
* severe chronic disease (cancer, IBD, malabsorption, malnutrition, chronic inflammatory diseases, renal, hepatic or cardiac diseases, COPD, respiratory insufficiency)
* chronic abdominal pain
* malformation of fingers
* systemic treatment or topical treatment likely to interfere with evaluation of the study parameters: antibiotics, intestinal or respiratory antiseptics, anti-rheumatics, antiphlogistics (except aspirin or equivalent products preventing from aggregation of platelets or blood clotting) and steroids prescribed in chronic inflammatory diseases
* other treatments likely to interfere with study outcome (e.g. laxatives, body weight management and/or medication)
* treatments with calcium antagonists and nitrates and alpha blockers
* diabetes mellitus on drug therapy
* severe neurological, cognitive or psychiatric diseases
* surgery or intervention requiring general anaesthesia within 2 months before the study
* vegetarian, vegan
* eating disorders (e.g. anorexia, bulimia)
* alcohol and drug abuse
* pregnancy or lactation
* legal incapacity
* blood parameters: Hb < 12 g/dL Liver transaminases (ALT, AST) > 2-fold increased Serum creatinine > 1,2 mg/dL

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Geometric mean titre of antibodies against one of the 3 influenza strains in HI test | 3 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, MD, Principal Investigator — Clinical Research Center Kiel GmbH